CLINICAL TRIAL: NCT04875676
Title: A Phase 1b, Open-label, Boost-optimization Study of an Adenoviral- Vector Based Oral Norovirus Vaccine (VXA-G1.1-NN) Expressing GI.1 VP1 Administered Orally to Healthy Adult Volunteers
Brief Title: Immunogenicity & Safety Study of Adenovirus Type 5 (AD5) Based Oral Norovirus Vaccines
Acronym: VXA-NVV-105
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VXA-NVV-105
Record Dates: First submitted 2021-04-19; First posted 2021-05-06 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Norovirus Infections
MeSH Terms: conditions — Caliciviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (4-week boost vaccination) (Active Comparator): (4-week boost vaccination) 10 subjects will receive two doses of 1x10 log10 IU ± 0.5 log at Day 1 and Week 4
  Interventions: Biological: VXA-G1.1-NN
- Cohort 2 (8-week boost vaccination) (Active Comparator): (8-week boost vaccination) 10 subjects will receive two doses of 1x10 log10 IU± 0.5 log at Day 1 and Week 8
  Interventions: Biological: VXA-G1.1-NN
- Cohort 3 (12-week boost vaccination) (Active Comparator): (12-week boost vaccination) 10 subjects will receive two doses of 1x10 log10 IU± 0.5 log at Day 1 and Week 12
  Interventions: Biological: VXA-G1.1-NN

INTERVENTIONS:
Biological: VXA-G1.1-NN — Norovirus GI.1 Norwalk VP1 Vaccine, Oral E1-/E3-Deleted Replication Defective Recombinant Adenovirus 5 with double-stranded RNA Adjuvant

SUMMARY:
To evaluate the immunogenicity of VXA-G1.1-NN with repeat-dose administration at Day 1 and varying boost schedules (Week 4, 8 or 12 post initial dose) in healthy adults aged 18-55, inclusive, and to assess the safety and tolerability of VXA- G1.1-NN with repeat-dose administration at varying boost schedules (Week 4, 8 or 12) in healthy adults aged 18-55, inclusive

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for this study, participants must meet all the following:

Age

1. 18 to 55 years old inclusive at the time of signing the Informed Consent Form (ICF).

   Type of Participants
2. General good health, without significant uncontrolled medical illness, based on medical history, physical examination, vital signs, and clinical laboratories (CBC, chemistry, and urinalysis) as determined by the investigator in consultation with the Research Monitor and Sponsor
3. Body mass index (BMI) between 17 and 35 kg/m2 at screening
4. Available for all planned visits and phone calls, and willing to complete all protocol- defined procedures and assessments (including ability and willingness to swallow multiple small enteric-coated tablets per study dose).

   Gender and Reproductive Considerations
5. Male or female participants Contraception use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   a. Female participants must provide a negative pregnancy test at each required visit and fulfill one of the following criteria:
   * At least 1 year post-menopausal (defined as amenorrhea for ≥12 consecutive months prior to Screening without an alternative medical cause).
   * Women under 60 years will need to verify post-menopausal status via a follicle-stimulating hormone (FSH) test if another option to prevent potential pregnancy will not be utilized for 30 days prior to baseline vaccination and until 60 days after the last vaccination.
   * Surgically sterile
   * Use of oral, implantable, transdermal or injectable contraceptives for 30 days prior to initial vaccination and until 60 days after the last vaccination. The form of contraception must be approved by the Investigator
   * A reliable form of contraception must be approved by the Investigator (e.g., double barrier method, Depo-Provera, intrauterine device, Norplant, oral contraceptives, contraceptive patches).
   * Not be sexually active (abstinent) or be in a relationship with partner who is sterile (must be discussed with site staff and documented).

   Informed Consent
6. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* The participants must be excluded from participating in the study if they meet any of the following:

Medical Conditions

1. Presence of significant uncontrolled medical or psychiatric illness (acute or chronic) including institution of new medical/surgical treatment or significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months of screening and reconfirmed at baseline
2. Cancer, or received treatment for cancer, within past 3 years (excluding basal cell carcinoma or squamous cell carcinoma)
3. Presence of immunosuppression or medical condition possibly associated with impaired immune responsiveness, including diabetes mellitus 1 and 2
4. History of irritable bowel disease or other inflammatory digestive or gastrointestinal condition that could affect the distribution/safety evaluation of an orally administered vaccine targeting the mucosa of the small intestine.

   Such conditions may include but are not limited to:
   1. Esophageal Motility Disorder
   2. Malignancy
   3. Malabsorption
   4. Pancreaticobiliary disorders
   5. Irritable bowel syndrome
   6. Inflammatory Bowel Disease
   7. Surgical Resection
   8. GERD
   9. Hiatal Hernia
   10. Peptic Ulcer (History of cholecystectomy is not exclusionary)
5. History of any form of angioedema
6. History of serious reactions to any vaccination such as anaphylaxis, respiratory problems, hives or abdominal pain
7. Diagnosed bleeding disorder or significant bruising or bleeding difficulties that could make blood draws problematic
8. Any condition that resulted in the absence or removal of the spleen
9. Acute disease within 72 hours prior to vaccination defined as the presence of a moderate or severe illness (as determined by the Investigator through medical history and physical exam). (Assessment may be repeated during screening period.)
10. Presence of a fever ≥ 38oC measured orally at baseline (Assessment may be repeated during screening period)
11. Any significant hospitalization within the last year which in the opinion of the Investigator or Sponsor could interfere with study participation.
12. Any other condition that in the clinical judgment of the investigator would jeopardize the safety or rights of a participant taking in the study, would render the participant unable to comply with the protocol or would interfere with the evaluation of the study endpoints Diagnostic Assessments
13. Positive human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) tests at the screening visit
14. Positive urine drug screen for drugs of abuse at screening
15. Positive breath or urine alcohol test at screening and baseline Prior/Concurrent Therapy
16. Receipt of a licensed vaccine within 14 days prior to baseline vaccination or planned administration during the study active period (4 weeks post each study vaccination).
17. Use of antibiotics, proton pump inhibitors, H2 blockers or antacids within 7 days prior to study drug administration or planned use during the active study period
18. Use of medications known to affect the immune function (e.g., systemic corticosteroids and others) within 2 weeks before study drug administration or planned use during the active study period
19. Daily use of nonsteroidal anti-inflammatory drugs within 7 days prior to study drug administration or planned use during the active study period
20. Administration of any investigational vaccine, drug or device within 8 weeks preceding study drug administration (Day 1), or planned use within the duration of the study Other Exclusions
21. Donation or use of blood or blood products within 30 days prior to study drug administration or planned donation during the active study period
22. History of drug, alcohol or chemical abuse within 1 year of screening
23. History of hypersensitivity or allergic reaction to any component of the investigational vaccine, including but not limited to fish gelatin

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Paguntalan, MD, Principal Investigator — Icon, Inc.
Locations (1):
- WCCT Global, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 (4-week Boost Vaccination) | Cohort 2 (8-week Boost Vaccination) | Cohort 3 (12-week Boost Vaccination)
Started | 10 | 10 | 10
Completed | 9 | 10 | 10
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (4-week Boost Vaccination) | Cohort 2 (8-week Boost Vaccination) | Cohort 3 (12-week Boost Vaccination) | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (7.42) | 35.4 (9.97) | 34.9 (10.09) | 37.8 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 4 | 15
  Male | 6 | 3 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 3 | 9
  Not Hispanic or Latino | 7 | 7 | 7 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 3 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 4
  White | 3 | 5 | 7 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30
Height [Mean (Standard Deviation); unit: centimeter] | 163.23 (7.236) | 175.63 (7.850) | 166.22 (10.734) | 168.36 (10.001)
Weight [Mean (Standard Deviation); unit: kilogram] | 75.22 (9.359) | 86.99 (20.457) | 75.54 (13.360) | 79.25 (15.603)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.27 (3.248) | 27.94 (4.940) | 27.32 (3.917) | 27.84 (3.971)
Vaccinated for COVID-19 [Count of Participants; unit: Participants]
  Yes - Pfizer-BioNTech | 4 | 3 | 3 | 10
  Yes - Moderna | 4 | 3 | 0 | 7
  Yes - Johnson & Johnson | 0 | 0 | 0 | 0
  Yes - Other | 0 | 0 | 0 | 0
  No | 2 | 4 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Viral-capsid Protein 1 (VP1)-Specific Antibody Secreting Cells (ASC) by Enzyme-linked Immunospot (ELISpot) Assay
Description: Comparison of VPI specific immunoglobin A (IgA) ASC levels between the 3 study cohorts by enzyme-linked immunospot (ELISpot) assay
Time Frame: Day 1 (Initial Vaccination) through Day 8 post boost (Second Vaccination)
Population: 1 subject received 1 dose only (8-week boost cohort)
Measure: Mean (95% Confidence Interval); unit: Spot Forming Units per 10^6 PBMC
Arm/Group | Cohort 1 (4-week Boost Vaccination) | Cohort 2 (8-week Boost Vaccination) | Cohort 3 (12-week Boost Vaccination)
Number analyzed (Participants) | 10 | 10 | 10
Spot Forming Units per 10^6 PBMC
  First Dose | 1.3 [-0.4 to 3.0] | 0.5 [-0.4 to 1.3] | 0.3 [-0.2 to 0.8]
  7-Days post First Dose | 127.6 [23.8 to 231.4] | 214.3 [15.8 to 412.9] | 327.5 [-106.4 to 761.4]
  Second Dose: number analyzed (Participants) | 10 | 9 | 10
  Second Dose | 2 [0.1 to 4.0] | 2.1 [-1.1 to 5.2] | 2.3 [-0.3 to 4.8]
  7-Days post Second Dose: number analyzed (Participants) | 10 | 9 | 10
  7-Days post Second Dose | 25.5 [-6.2 to 57.2] | 68.8 [-29.4 to 167.0] | 132.1 [-16.1 to 280.4]

2. Primary Outcome: Norovirus G1.1 Histo-blood Group Antigen (HBGA) Blocking Antibodies (BT50) Assay
Description: Comparison of subjects with a ≥2-, 3- or 4-fold increase over baseline titer of GI.1 histo-blood group antigen (HBGA) blocking antibodies (BT50) levels between the 3 study cohorts.
Time Frame: Day 1 (Initial Vaccination) through Day 29 post boost (Second Vaccination)
Population: 1 subject received 1 dose only (8-week boost cohort)
Measure: Geometric Mean (95% Confidence Interval); unit: 10^6 AU/mL
Arm/Group | Cohort 1 (4-week Boost Vaccination) | Cohort 2 (8-week Boost Vaccination) | Cohort 3 (12-week Boost Vaccination)
Number analyzed (Participants) | 10 | 10 | 10
10^6 AU/mL
  Day of First Dose: GMC (geometric mean concentration) | 29.9 [17.0 to 52.6] | 27.9 [12.8 to 60.9] | 21.1 [12.0 to 37.1]
  28-Days post First Dose: GMC (geometric mean concentration) | 52.7 [28.8 to 96.2] | 69.5 [23.2 to 208.4] | 54.9 [18.7 to 161.2]
  28-Days post Second Dose: GMC (geometric mean concentration): number analyzed (Participants) | 10 | 9 | 10
  28-Days post Second Dose: GMC (geometric mean concentration) | 74.5 [36.9 to 150.4] | 54.0 [19.0 to 153.8] | 64.9 [24.4 to 172.8]

3. Primary Outcome: VP1 Serum Immunoglobin G (IgG) by Mesoscale Discovery (MSD) Assay
Description: Comparison of VPI specific immunoglobin A (IgA) ASC levels by Mesoscale Discovery (MSD) assay between the 3 study cohorts
Time Frame: Day 1 (Initial Vaccination) through Day 29 post boost (Second Vaccination)
Population: 1 subject received 1 dose only (8-week boost cohort)
Measure: Geometric Mean (95% Confidence Interval); unit: 10^6 AU/mL
Arm/Group | Cohort 1 (4-week Boost Vaccination) | Cohort 2 (8-week Boost Vaccination) | Cohort 3 (12-week Boost Vaccination)
Number analyzed (Participants) | 10 | 10 | 10
10^6 AU/mL
  First Dose: GMC (geometric mean concentration) | 0.5 [0.1 to 2.1] | 0.3 [0.1 to 1.2] | 0.2 [0.0 to 1.1]
  28-Days post the First Dose: GMC (geometric mean concentration) | 2.1 [0.9 to 4.9] | 2.6 [0.8 to 8.7] | 2.1 [0.4 to 11.2]
  28-Days post the Second Dose: GMC (geometric mean concentration): number analyzed (Participants) | 10 | 9 | 10
  28-Days post the Second Dose: GMC (geometric mean concentration) | 1.5 [0.6 to 3.9] | 1.2 [0.4 to 3.6] | 1.7 [0.5 to 6.1]

4. Primary Outcome: Norovirus G1.1 Histo-blood Group Antigen (HBGA) Blocking Antibodies (BT50) Assay
Description: Comparison of GI.1 histo-blood group antigen (HBGA) blocking antibodies (BT50) levels between the 3 study cohorts
Time Frame: Day 1 (Initial Vaccination) through Day 29 post boost (Second Vaccination)
Population: 1 subject received 1 dose only (8-week boost cohort)
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Cohort 1 (4-week Boost Vaccination) | Cohort 2 (8-week Boost Vaccination) | Cohort 3 (12-week Boost Vaccination)
Number analyzed (Participants) | 10 | 10 | 10
Fold Rise
  28-Days post First Dose: GMFR (geometric mean fold rise) | 1.8 [1.2 to 2.7] | 2.5 [1.2 to 5.4] | 2.6 [1.3 to 5.1]
  28-Days post Second Dose: GMFR (geometric mean fold rise) | 2.5 [1.5 to 4.1] | 2.4 [1.3 to 4.3] | 3.1 [1.8 to 5.1]

5. Secondary Outcome: Solicited Symptoms of Reactogenicity
Description: Comparison of frequency, duration, and severity of solicited symptom events in participants
Time Frame: Day 1 (Vaccination) to Day 8 post each vaccination
Population: Subjects with Solicited Symptoms
Measure: Number; unit: events
Arm/Group | Cohort 1 (4-week Boost Vaccination) | Cohort 2 (8-week Boost Vaccination) | Cohort 3 (12-week Boost Vaccination)
Number analyzed (Participants) | 10 | 10 | 10
events
  Fever: Total | 0 | 0 | 0
  Fever: Mild | 0 | 0 | 0
  Fever: Moderate | 0 | 0 | 0
  Headache: Total | 5 | 1 | 5
  Headache: Mild | 4 | 1 | 3
  Headache: Moderate | 1 | 0 | 2
  Myalgia: Total | 2 | 1 | 2
  Myalgia: Mild | 2 | 0 | 2
  Myalgi: Moderate | 0 | 1 | 0
  Abdominal Pain: Total | 2 | 2 | 3
  Abdominal Pain: Mild | 2 | 1 | 2
  Abdominal Pain: Moderate | 0 | 1 | 1
  Anorexia: Total | 1 | 0 | 0
  Anorexia: Mild | 1 | 0 | 0
  Anorexia: Moderate | 0 | 0 | 0
  Nausea: Total | 1 | 0 | 2
  Nausea: Mild | 1 | 0 | 2
  Nausea: Moderate | 0 | 0 | 0
  Vomiting: Total | 1 | 0 | 2
  Vomiting: Mild | 1 | 0 | 2
  Vomiting: Moderate | 0 | 0 | 0
  Diarrhea: Total | 3 | 2 | 4
  Diarrhea: Mild | 2 | 1 | 3
  Diarrhea: Moderate | 1 | 1 | 1
  Malaise/Fatigue: Total | 3 | 1 | 3
  Malaise/Fatigue: Mild | 2 | 1 | 2
  Malaise/Fatigue: Moderate | 1 | 0 | 1

6. Other Pre Specified Outcome: Unsolicited Adverse Events (AEs)
Description: Comparison of the frequency, duration, and severity of unsolicited AEs and serious AEs (SAEs) including AEs of Special Interest (AESIs) and new onsets of chronic illness (NOCIs) in participants
Time Frame: Day 1 (Vaccine) through 28 days following boost (Second Vaccination)
Population: Subjects with Any Unsolicited AEs
Measure: Number; unit: events
Arm/Group | Cohort 1 (4-week Boost Vaccination) | Cohort 2 (8-week Boost Vaccination) | Cohort 3 (12-week Boost Vaccination)
Number analyzed (Participants) | 10 | 10 | 10
events
  Syncope (Mild) | 1 | 0 | 1
  Toothache (Mild) | 0 | 0 | 1
  COVID-19 Pneumonia (Severe) | 0 | 1 | 0

7. Other Pre Specified Outcome: Long-term Safety
Description: Frequency, duration, and severity of all SAEs, AESIs and NOCIs through 6 months after last vaccination.
Time Frame: Day 1 (Vaccine) through 6 months following boost (Second Vaccination)
Reporting Status: Not Posted

8. Primary Outcome: VP1 Serum Immunoglobin G (IgG) by Mesoscale Discovery (MSD) Assay
Description: as for outcome 3
Time Frame: Day 1 (Initial Vaccination) through Day 29 post boost (Second Vaccination)
Population: 1 subject received 1 dose only (8-week boost cohort)
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Cohort 1 (4-week Boost Vaccination) | Cohort 2 (8-week Boost Vaccination) | Cohort 3 (12-week Boost Vaccination)
Number analyzed (Participants) | 10 | 10 | 10
Fold rise
  28-Days post the First Dose: GMFR (geometric mean fold rise) | 4.6 [1.6 to 13.6] | 8.9 [3.9 to 20.5] | 11.3 [3.4 to 37.0]
  28-Days post the Second Dose: GMFR (geometric mean fold rise) | 3.3 [1.3 to 8.5] | 5.4 [2.5 to 11.7] | 8.9 [2.9 to 26.8]

ADVERSE EVENTS:
Time Frame: 6 months following boost dose
Description: AEs were categorized by solicited AEs, unsolicited AEs (including both AESIs and NOCIs), and SAEs, where the frequencies and durations of each were summarized by cohort, severity, and relatedness to study treatment.
Arm/Group | Cohort 1 (4-week Boost Vaccination) | Cohort 2 (8-week Boost Vaccination) | Cohort 3 (12-week Boost Vaccination)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 3/10 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (4-week Boost Vaccination) (N=10) | Cohort 2 (8-week Boost Vaccination) (N=10) | Cohort 3 (12-week Boost Vaccination) (N=10)
COVID-19 Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hospitalization (Investigations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (4-week Boost Vaccination) (N=10) | Cohort 2 (8-week Boost Vaccination) (N=10) | Cohort 3 (12-week Boost Vaccination) (N=10)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) — Fever
Headache (Nervous system disorders) | 5 (5) | 1 (1) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4)
Fatigue (General disorders) | 3 (3) | 1 (1) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT04875676/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT04875676/SAP_001.pdf